CLINICAL TRIAL: NCT01039922
Title: SwissNET - a Prospective Registry of Patients With Neuroendocrine Tumours in Switzerland
Brief Title: SwissNET - a Registry for Neuroendocrine Tumours in Switzerland
Acronym: SwissNET
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); University Hospital, Basel, Switzerland (Other); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other); University Hospital, Zürich (Other); Triemlispital Zurich (Unknown); Spitalnetz Bern (Unknown); Ente Ospedaliero Cantonale, Bellinzona (Other); Luzerner Kantonsspital (Other); Kantonsspital Liestal (Other); Kantonsspital Graubuenden (Other); Spital Limmattal Schlieren (Other); Waid City Hospital, Zurich (Other); Spital STS AG (Industry)
Responsible Party: Sponsor
Other Study IDs: BAG 035.0002-20/19; 395/2014 (Other: KEK)
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumor
Keywords: Neuroendocrine Tumors; Registries
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with a histologically confirmed diagnosis of a neuroendocrine tumor irrespective of primary tumor location

SUMMARY:
Gastroentero-pancreatic neuroendocrine tumours (GEP-NETs) are regarded as a fairly rare disease. They are derived from the neuroendocrine system of the gastrointestinal tract and the pancreas and share common clinical features. So far, there is still uncertainty about the cell biology and mechanistic regulation of these tumours. Therefore targeted treatment is limited and management challenging. Treatment options include surgery, medical and ablative therapy, and more recently peptide-receptor radionuclide therapy. In order to better understand the characteristics of GEP-NETs and to evaluate treatment strategies, the SwissNET registry aims at the collection of data from patients presenting with a GEP-NET in Switzerland. Data will be entered prospectively and anonymized in a specifically designed database after the patient has given informed consent. All hospitals and general practitioners are invited to report on patients with a GEP-NET diagnosis and to participate to the registry. Data will be evaluated within regular time frames, focussing on types of GEP-NETs, treatment modalities and patient outcomes (e.g. mortality, hospitalisation rate), thereby contributing to the better understanding of these tumours.

DETAILED DESCRIPTION:
Background

Gastroentero-pancreatic neuroendocrine tumours (GEP-NETs) are generally classified as rare diseases. Little is known about their cell biology and their mechanistic regulation. During the last years, the incidence of GEP-NETs is continuously increasing worldwide. In parallel, novel treatment options are currently evaluated which may substantially improve prognosis of patients with NETs. Data on such tumours in Switzerland, however, is scarce and treatment strategies vary throughout the country.

Objective

To systematically and prospectively collect clinical information of patients with GEP-NETs in Switzerland based on a histologically confirmed diagnosis.

Methods

All NETs of both, gastrointestinal and pulmonary origin are included provided that patients have given informed consent. Data will be entered prospectively and anonymised in a specifically designed database. Contributing centres and general practitioners are visited by a study nurse, patient files are analysed and data is transferred to the database. In case of conflicting evidence, questions are resolved in collaboration with a review board of SwissNET. Evaluation of treatment modalities and patient outcomes (e.g. mortality, hospitalisation rate) will take place within regular time frames.

ELIGIBILITY:
Inclusion Criteria:

* Neuroendocrine tumor irrespective of primary tumor location
* Diagnosis in Switzerland
* Given informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected either through the report of a pathological institute or of any medical doctor within Switzerland treating patients with neuroendocrine tumours.
Sampling Method: Non-Probability Sample
Enrollment: 1245 (Estimated)
Dates: Start 2008-01; Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Tumor-related mortality | Every 5 years

SECONDARY OUTCOMES:
Incidence of GEP-NET in Switzerland | Every 5 years
Effect of specific treatment strategies | Every 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aurel Perren, MD, Study Director — Institute of Pathology, University of Bern, Bern
Locations (55):
- Switzerland (55):
  - Kantonsspital Aarau, Aarau
  - Spitalnetz Bern Aarberg, Aarberg
  - Bezirksspital Affoltern, Affoltern am Albis
  - Kantonsspital Uri, Altdorf, Altdorf
  - St. Claraspital, Basel
  - Universitätsspital Basel, Basel
  - Istituto oncologico della Svizzera italiana, Bellinzona
  - Div. of Endocrinology, Diabetes and Clinical Nutrition, Bern University Hospital, Bern
  - Spital Tiefenau, Spitalnetz Bern, Bern
  - Zieglerspital Bern, Bern
  - Spitalzentrum Biel - Bienne, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - Regionsspital Emmental, Burgdorf
  - Kantonsspital Chur, Chur
  - Private practise Dr. Mannhart, Churwalden
  - Hôpital du Jura, Delémont
  - Spital Dornach, Dornach
  - Regionalspital Einsiedeln, Einsiedeln
  - Hôpitaux Universitaires de Genève, Geneva
  - Spital Grabs, Grabs
  - See-Spital Horgen, Horgen
  - Spital Zimmerberg, Horgen
  - Fmi Spital Interlaken, Interlaken
  - Spital Lachen, Lachen
  - Spital Region Oberaargau, Langenthal
  - Kantonsspital Laufen, Laufen
  - Centre hospitalier universitaire vaudois, CHUV, Lausanne
  - Kantonsspital Liestal, Liestal
  - Hirslandenklinik St. Anna, Lucerne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Sursee, Luzern, Lucerne
  - Kreisspital Männedorf, Männedorf
  - Kantonsspital Münsterlingen, Münsterlingen
  - Kantonsspital Olten, Olten
  - Gesundheitszentrum Fricktal, Rheinfelden
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Obwalden, Sarnen
  - Spital Limmattal, Schlieren
  - Spital Schwyz, Schwyz
  - Privatpraxis Dr. H.J. Poths, Seuzach Dorf
  - Centre hospitalier du centre du Valais, Sion
  - Bürgerspital Solothurn, Solothurn
  - Kantonsspital Nidwalden, Stans
  - Thun Spital STS AG, Thun
  - Spital Uster, Uster
  - Regionalspital Visp, Visp
  - Kantonsspital Winterthur, Winterthur
  - Kantonsspital Wolhusen, Wolhusen
  - Spital Zollikerberg, Zollikerberg
  - Zuger Kantonsspital AG, Zug
  - Pathologie Medica Zürich, Zurich
  - Stadtspital Triemli, Zurich
  - Stadtspital Waid, Zurich
  - Universitätsspital Zürich, Zurich
  - STS AG Spital Zweisimmen, Zweisimmen